CLINICAL TRIAL: NCT01267175
Title: United Kingdom User Evaluation, MiniMed Paradigm® X54 System
Acronym: X54User
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Scott Lee, MD, Medtronic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ETP08-2625
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- X54 pump (Experimental): All subjects transferred from current pump to X54
  Interventions: Device: X54 insulin pump with low suspend feature

INTERVENTIONS:
Device: X54 insulin pump with low suspend feature — Change from current insulin pump to new X54 pump
  Other Names: Veo

SUMMARY:
The user evaluation is to assess user acceptance and the quality of training materials for the MiniMed Paradigm® X54 System (X54 System) in preparation for commercial distribution of the new system.

ELIGIBILITY:
Inclusion Criteria:

* Are current 512/712, 515/715 or 522/722 MiniMed Paradigm Insulin Pump users, with or without CGM experience, and have at least three months experience with any one of these devices;
* Have signed an Informed Consent and are willing to comply with the user evaluation procedures;
* Have an HbA1c value less than 9.0% recorded at the time of their last test (if no HbA1c value is available within three months of enrollment, an HbA1c should be performed prior to entry to verify inclusion criteria);
* Are willing to use the Bolus Wizard feature;
* Agree to complete a diary for the duration of the study;
* Agree to complete a questionnaire at the conclusion of the study;
* Have been diagnosed with Type 1 Diabetes Mellitus by appropriate fasting or non fasting lab blood glucose values, c-peptide, insulin antibodies, prior documented DKA or good clinical picture at least six months prior to study start;
* Are 18 - 65 years of age;
* Have access to the internet and agree to upload the device per protocol

Exclusion Criteria:

* Is pregnant or planning to become pregnant during the course of the user evaluation. Pregnancy screening will be completed during the routine office visit prior to evaluation for the study. If a woman becomes pregnant during participation, she will be withdrawn;
* Suffers from a chronic debilitating condition;
* Has serious or unstable medical or psychological conditions (e.g., eating disorders, clinical depression, anxiety disorder) which, in the opinion of the Investigator, would compromise the subject's safety or successful participation in the study;
* Has impaired vision or hearing problems that could compromise the handling of the device;
* Has a history of tape allergies or skin conditions that could interfere with continued use of the system;
* Has the potential for lack of compliance or any other issue, in the opinion of the Investigator, that may preclude the subject from satisfactory participation in the study;
* Has travel plans which would make it difficult for the subject to attend on-site study visits as scheduled;
* Is currently participating in an investigational study (drug or device).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Lee, MD, Study Director — Medtronic
Locations (6):
- United Kingdom (6):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Kings College Hospital, Denmark Hill, London
  - Harrogate District Hospital, Harrogate, N. Yorkshire
  - Newcastle General Hospital, Newcastle upon Tyne, Tyne and Wear
  - Guy's Hospital, London

REFERENCES:
- [Derived] Choudhary P, Shin J, Wang Y, Evans ML, Hammond PJ, Kerr D, Shaw JA, Pickup JC, Amiel SA. Insulin pump therapy with automated insulin suspension in response to hypoglycemia: reduction in nocturnal hypoglycemia in those at greatest risk. Diabetes Care. 2011 Sep;34(9):2023-5. doi: 10.2337/dc10-2411. PMID 21868778

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | X54 Pump
Started | 31
Completed | 29
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | X54 Pump
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 31

OUTCOME MEASURES:

1. Primary Outcome: Usability of the X54 Insulin Pump Meets Expectations
Description: Questionnaire completed at the end of the study measuring usability of the X54 insulin pump. Results scored on a Likert scale of 1 - 7, 1 being the least likely to use and 7 being the most likely to use.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | X54 Pump
Number analyzed (Participants) | 31
Scores on a scale | 5.9 (1.56)

2. Secondary Outcome: Usability of the Training Material Meets Expectations
Description: Questionnaire completed at the end of the study, measuring usability of the device training manual. Results scored on a Likert scale of 1 - 7, 1 being the least user friendly and 7 being the most user friendly.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | X54 Pump
Number analyzed (Participants) | 31
Scores on a scale | 6.1 (1.16)

ADVERSE EVENTS:
Time Frame: Unanticipated Device related Adverse Events were required to be reported over the 15 week observation period.
Arm/Group | X54 Pump
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days